CLINICAL TRIAL: NCT04005859
Title: Pain Control in Colorectal Surgery: Liposomal Bupivacaine Block Versus Intravenous Lidociane
Acronym: Exparel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01-18-16
Record Dates: First submitted 2019-06-27; First posted 2019-07-02 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2021-10

CONDITIONS: Colorectal Disorders
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTROL: IV Lido (Active Comparator): CONTROL: Intravenous lidocaine, pre- and post-surgery (IV Lido)
  Interventions: Drug: IV Lidocaine
- EXPERIMENTAL: Exparel (Experimental): EXPERIMENTAL: TAP block with liposomal bupivacaine will be given as an injection (Exparel)
  Interventions: Drug: Exparel

INTERVENTIONS:
Drug: Exparel — 2. Liposomal bupivacaine TAP block (experimental arm)
  1. Block will be administered after induction of anesthesia and before incision by a specifically trained attending surgeon or surgical fellow with the colorectal service.
  2. A single vial of liposomal bupivacaine (20 mL 1.3%, 13.3mg/mL, 266 mg) will be diluted in 50cc bupivacaine to a volume of 60cc prior to administration. This will be divided into 2 doses for bilateral TAP blocks.
  3. The LB will be administered under ultrasound guidance in the transversus abdominis plain per manufacturer recommendations.
  4. Adhesive tapes will be applied at the level of the TAP block puncture sites.
  Arms: EXPERIMENTAL: Exparel
Drug: IV Lidocaine — 1. Intravenous Lidocaine infusion (control arm, current standard of care)
  1. 100 mg/5mL intravenous bolus of lidocaine 2% PF 5mL will be initiated by anesthesia service prior to general anesthesia induction.
  2. 1.5 mg/kg/hr to begin prior to incision and continue until discontinued 1 hr postoperatively in PACU. Patients will be monitored in PACU for at least 30 minutes after discontinuation of lidocaine drip.
  3. Adhesive tapes will be applied at the presumed level of TAP block puncture sites.
  Arms: CONTROL: IV Lido

SUMMARY:
To compare the analgesic impact of intravenous perioperative lidocaine infusion with preoperative liposomal bupivacaine TAP block in colorectal surgery. This is to be integrated into the standard ERAS protocol currently utilized at Carolinas Medical Center. Primary endpoints will be postoperative pain as measured by verbal rate scale (VRS), postoperative morphine equivalents utilized per day, and over 30 days. Secondary endpoints will include date of ambulation, return of bowel function (first flatus), tolerance of goal diet, incidence of post-operative nausea and vomiting during hospital stay, length of stay (hospital and PACU), post-operative morbidity (Clavien-Dindo, related to both anesthesia and surgery), cost of hospitalization (operative, PACU, postoperative stay, and total) and quality of life on follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Elective laparoscopic colorectal surgery
* ASA I-III

Exclusion Criteria:

* Contraindication to Na Channel Blocker
* Chronic Opioid use
* Liver dysfunction
* Renal insufficiency
* Epilepsy
* Psychomotor retardation
* BMI >40
* Sleep Apnea
* Cardiac Rhythm Disorders
* Planned open or concomitant procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2021-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kasten, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health - Carolinas Medical Center, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CONTROL: IV Lido: CONTROL: Intravenous lidocaine, pre- and post-surgery (IV Lido)
  IV Lidocaine: 1. Intravenous Lidocaine infusion (control arm, current standard of care) n= 35
  1. 100 mg/5mL intravenous bolus of lidocaine 2% PF 5mL will be initiated by anesthesia service prior to general anesthesia induction.
  2. 1.5 mg/kg/hr to begin prior to incision and continue until discontinued 1 hr postoperatively in PACU. Patients will be monitored in PACU for at least 30 minutes after discontinuation of lidocaine drip.
  3. Adhesive tapes will be applied at the presumed level of TAP block puncture sites.
- EXPERIMENTAL: Exparel: EXPERIMENTAL: TAP block with liposomal bupivacaine will be given as an injection (Exparel)
  Exparel: 2. Liposomal bupivacaine TAP block (experimental arm) n= 35
  1. Block will be administered after induction of anesthesia and before incision by a specifically trained attending surgeon or surgical fellow with the colorectal service.
  2. A single vial of liposomal bupivacaine (20 mL 1.3%, 13.3mg/mL, 266 mg) will be diluted in 50cc bupivacaine to a volume of 60cc prior to administration. This will be divided into 2 doses for bilateral TAP blocks.
  3. The LB will be administered under ultrasound guidance in the transversus abdominis plain per manufacturer recommendations.
  4. Adhesive tapes will be applied at the level of the TAP block puncture sites.
Period: Overall Study
Arm/Group | CONTROL: IV Lido | EXPERIMENTAL: Exparel
Started | 32 | 29
Completed | 28 | 25
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CONTROL: IV Lido | EXPERIMENTAL: Exparel | Total
Number analyzed (Participants) | 28 | 25 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (16.2) | 55.8 (14) | 55.4 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 25
  Male | 19 | 9 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.7 (5.3) | 29.6 (8.2) | 28.4 (7.0)
On Steroids [Count of Participants; unit: Participants] | 4 | 1 | 5
H/O Diabetes [Count of Participants; unit: Participants] | 3 | 6 | 9
Current Tobacco Use [Count of Participants; unit: Participants] | 7 | 6 | 13
Prior intra-abdominal surgery [Count of Participants; unit: Participants] | 5 | 9 | 14
Procedure was robotic-assisted [Count of Participants; unit: Participants] | 14 | 9 | 23

OUTCOME MEASURES:

1. Primary Outcome: Verbal Pain Scale (VRS) - 4 Week Post-op
Description: Postoperative pain was measured by verbal rate scale (VRS) Scale of 0-10 at instance of 4-week post-op visit (or phone call). 0 represents no pain while 10 represents worst possible pain.
Time Frame: Single VRS assessed at 4-week post-op visit (or phone call)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CONTROL: IV Lido | EXPERIMENTAL: Exparel
Number analyzed (Participants) | 28 | 25
score on a scale | 0.4 (0.7) | 1.1 (2.0)

ADVERSE EVENTS:
Time Frame: 4 weeks from date of surgery (scheduled time of post-op clinic visit addressing primary endpoint of total OME utilized by patient)
Arm/Group | CONTROL: IV Lido | EXPERIMENTAL: Exparel
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/25
Other Adverse Events (participants affected / at risk) | 0/28 | 0/25

LIMITATIONS AND CAVEATS:
1. Opioid consumption was quite varied amongst patients, possibly contributing to underpowered study.
2. Inconsistent recording of VAS while inpatient
3. Inconsistent recording of VAS while undergoing 2 and 4 week post-op follow-up (clinic vs phone)
4. Difficult to completely account for OME based on potential for outside prescriptions not seen by researchers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT04005859/Prot_SAP_001.pdf
  • Informed Consent Form (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT04005859/ICF_002.pdf